CLINICAL TRIAL: NCT02112474
Title: The Pain Suppressive Effect of Low Frequency Spinal Cord Stimulation Versus High Frequency Spinal Cord Stimulation
Brief Title: The Pain Suppressive Effect of Alternative Spinal Cord Stimulation Frequencies
Acronym: HALO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Breel (Other)
Collaborators: Diakonessenhuis, Utrecht (Other); Rijnstate Hospital (Other); Alrijne Hospital (Other); Noordwest Ziekenhuisgroep (Other)
Responsible Party: Sponsor-Investigator, Jennifer Breel, Study Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MDT-HF-2013; NL43067.018.13 (Other: CCMO); 2013_281 (Other: METC Academic_Medical _Center)
Record Dates: First submitted 2014-03-25; First posted 2014-04-14 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Failed Back Surgery Syndrome; Neuropathic Pain
Keywords: Failed Back Surgery Syndrome; Neuropathic pain; Leg Pain; Chronic Pain; Spinal Cord Stimulation; Neurostimulation
MeSH Terms: conditions — Failed Back Surgery Syndrome; Neuralgia; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Cord Stimulation Group 1 (Experimental): 9 days of spinal cord stimulation at 30 Hertz and perceptible paraesthesias
  Interventions: Device: Spinal Cord Stimulation; Device: Group 1
- Spinal Cord Stimulation Group 2 (Experimental): 9 days of spinal cord stimulation with 1000 Hertz and sub-perception paraesthesias
  Interventions: Device: Spinal Cord Stimulation; Device: Group 2

INTERVENTIONS:
Device: Spinal Cord Stimulation — Crossover design whereby subjects will undergo Spinal Cord Stimulation in two arms: low frequency stimulation and high frequency stimulation
Device: Group 1 — 9 days of spinal cord stimulation at 30 Hertz and perceptible paraesthesias
  Arms: Spinal Cord Stimulation Group 1
Device: Group 2 — 9 days of spinal cord stimulation with 1000 Hertz and sub-perception paraesthesias
  Arms: Spinal Cord Stimulation Group 2

SUMMARY:
Electrical stimulation of the spinal cord (Spinal Cord Stimulation or SCS) for pain relief has been used for decades. It is used most commonly in patients with chronic neuropathic leg pain, after spinal surgery. Conventional neurostimulation is applied in frequencies of 30 to 60 Hertz (Hz) and perceptible paraesthesias are felt. Stimulation using higher frequencies with sub perception paraesthesias has recently challenged the conventional form of neurostimulation.The high frequency stimulation appears to show better pain relief for both back and limb pain in comparison to low frequency SCS, and may also to be effective in some subjects who did not respond to low frequency SCS.

DETAILED DESCRIPTION:
Rationale:

Electrical stimulation of the dorsal columns of the spinal cord (Spinal Cord Stimulation or SCS) for pain relief has been used in humans for several decades. The most common indication for SCS is the treatment of refractory neuropathic leg pain, particularly when these symptoms persist after an anatomically successful operation (Failed Back Surgery Syndrome or FBSS).

Low frequency - conventional - SCS (LF-SCS) is applied in frequencies ranging from 30 to 60 Hertz (Hz) and the subject feels paraesthesias in the painful area, which is considered the ideal situation. Recently, LF-SCS has been challenged by the development of stimulation modes at higher frequencies which provide pain relief at sub-perception threshold, i.e. without paraesthesias. A recent case series reported that High Frequency Spinal Cord Stimulation (HF-SCS) appears to show better pain relief for both back and limb pain in comparison to LF-SCS, and also to be effective in some subjects who did not respond to LF-SCS.

Objective:

The primary objective of this trial is to compare pain suppression in two groups of subjects with chronic unilateral limb pain as a result of FBSS .

Study design:

A prospective, double blind (subject, physician, statistician), multi-centre, randomized, crossover trial of SCS in the treatment of subjects with refractory neuropathic leg pain after back surgery.

Study population:

Patients with chronic neuropathic refractory unilateral leg pain

Intervention:

Patients will undergo neurostimulation with low and high frequency parameters, the order in which they receive treatment will be randomized

Main study endpoint:

Pain suppression in the short and long-term (24 days and 12 months)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Both methods of stimulation are standard clinical practice performed routinely in the study centres, both groups will receive this standard care. The only difference is change of stimulation frequency and the order in which it is applied.

Possible benefit to the subject is that both forms of stimulation will be evaluated. This may lead to a better quality of life in the HF-SCS Group as result of pain relief without paraesthesias. Furthermore, non-responders to LF-SCS may benefit from HF-SCS.

ELIGIBILITY:
Inclusion Criteria:

* Male/female, 18 years to 70 years
* Chronic, persistent, refractory, unilateral neuropathic limb pain, as a result of spinal surgery
* Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and minimally interventional pain procedures for chronic pain
* Pain radiating in the leg, following segments L4 and/or L5 and/or S1 for at least 6 months
* Minimum baseline pain intensity as assessed by VAS of ≥ 50mm on 100mm scale in the primary pain area
* Subject is able and willing to provide informed consent
* Subject is able and willing to comply with the protocol and follow-up schedule
* Subject has been included for implantation according to standard criteria from the Dutch Neuromodulation Society

Exclusion Criteria:

* Back pain component of more than 20% or VAS > 40mm on 100mm scale
* Bilateral limb pain
* Subjects with a previous SCS implantation.
* Changes in pain medication in the 2 months preceding the trial period;
* Expected inability of subjects to correctly operate the neurostimulation system
* Presence of any other clinically significant or disabling chronic pain condition -eg. hip arthrosis, rheumatoid arthritis, fibromyalgia, etc.
* History of coagulation disorders, lupus erythematosus, diabetes mellitus, or morbus Bechterew
* Symptoms or proof of any malignant disease
* Current use of medicines affecting coagulation which cannot be temporarily stopped
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* Life expectancy of less than 1 year
* Existing or planned pregnancy in the trial period
* BMI >20 and <35 - a minimum and maximum BMI limit are imposed due to the technical difficulties and risk of complications in underweight or morbidly obese subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scores (VAS) | 24 days
  0mm to 10mm line scale, where higher score is better, measured 4 times a day at 09:00, 15:00, 21:00 and a nightscore measured first thing in the morning

SECONDARY OUTCOMES:
Visual Analog Pain scores (VAS) | 12 months
  0mm to 10mm line scale, where higher score is better, measured 4 times a day at 09:00, 15:00, 21:00 and a nightscore measured first thing in the morning
EuroQoL 5Dimensions-3Levels | 1 month, 12 months
  Quality of LIfe, 5 questions measured on 3 levels (mild =1, moderate=2, severe=3). Higher score is worse. Each domain calculated according to a national index.
Short Form-36 | 1 month, 12 months
  Quality of Life, 36 questions with differing formats, 8 domains, higher score is better
Sleep questionnaire | 1 month, 12 months
  Quality of sleep before and after stimulation, Several Likert-type items 0-5 and 0-7, higher score is better
GPES | 1 month, 12 months
  Subject satisfaction,1 Likert-type item 0-7, higher score is better
Employment status | 12 months
  Change in employment status, open question whether or not employment status has changed and how many hours per week persons were/not working
(Serious) Adverse Events | 12 months
  Number of patients with device related events such as lead dislocation, infections, pocket pain, increase in pain whilst using one paticular frequency etc.

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Frank Wille, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jennifer S Breel, MPA,MSc., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Velp, Gelderland
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Alrijne Hospital, Leiderdorp, South Holland
  - Diakonessenhuis, Zeist, Utrecht

REFERENCES:
- [Derived] Breel J, Wille F, Wensing AGCL, Kallewaard JW, Pelleboer H, Zuidema X, Burger K, de Graaf S, Hollmann MW. A Comparison of 1000 Hz to 30 Hz Spinal Cord Stimulation Strategies in Patients with Unilateral Neuropathic Leg Pain Due to Failed Back Surgery Syndrome: A Multicenter, Randomized, Double-Blinded, Crossover Clinical Study (HALO). Pain Ther. 2021 Dec;10(2):1189-1202. doi: 10.1007/s40122-021-00268-7. Epub 2021 Jun 6. PMID 34091818